CLINICAL TRIAL: NCT01360099
Title: Bisphosphonate Users Radiographic Characteristics of the Hip (BURCH) Study
Status: Completed | Type: Observational
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 110156; 11-AR-0156
Record Dates: First submitted 2011-05-20; First posted 2011-05-25 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-01-11

CONDITIONS: Osteoporosis; Bone Diseases, Metabolic; Hip Fractures
Keywords: Atypical Hip Fracture; Biosphosphonates; Subtrochanteric Hip Fracture; Osteoporosis
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic; Hip Fractures

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- Osteoporosis is a condition where the bone becomes more brittle and more likely to break as a person ages. The drugs that people take to treat this condition have prevented many common hip fractures. But these drugs may be associated with problems in the shape and structure of the hip bone after many years of use. These changes in the hip bone may lead to an unusual kind of hip fracture. These fractures are very rare, so it is hard to study them. Researchers want to learn more about these fractures.

Objectives:

- To compare hip x-rays of three groups: people who have been taking osteoporosis drugs for several years, those who have just started taking them, and those who have never taken these drugs.

Eligibility:

* People at least 50 years of age who have been taking osteoporosis drugs for at least 5 years.
* People at least 50 years of age who have been taking these drugs for less than 1 year.
* People at least 50 years of age who have never taken these drugs.

Design:

* All participants will have three total visits over 3 years.
* At the first visit, those taking part will have a medical history and physical exam. They will complete a questionnaire about medication use and bone health. They will also have an x-ray of the hips and pelvis, and have a bone density scan (the kind used to test for osteoporosis) of the hips.

Those in the study will repeat these exams and medical history questions at followup visits. These visits will take place 18 months and 36 months after the first study visit.

* At any of these visits, participants who may have a hip fracture that does not show up on the x-rays will have an imaging study to examine the bone more closely.
* Participants who receive a hip replacement or suffer from a broken bone at any time should inform the study researchers as soon as possible.

DETAILED DESCRIPTION:
Objective:

Bisphosphonates are a class of medications that treat osteoporosis and prevent fractures, and have been available for more than a decade. However, there have been recent studies that have shown that, on rare occasions, they may be associated with an atypical hip fracture after long-term use. Radiographic features such as beaking and thickening along the side of the hip bone have been frequently observed with these atypical femur fractures, but most of the studies to date have only been focused on finding the fractures, not the x-ray features. It is not known how common these x-ray features and pain symptoms are amongst bisphosphonate users that have not yet experienced a fracture. If there is a difference between users and non-users, these features may be a valuable finding to help catch fractures before they happen. A recent hypothesis has emerged that a genetic condition, hypophosphatasia, may play a role.

Study population:

This study will evaluate the presence of these features in users of bisphosphonates and the general population. Individuals from the community who have taken bisphosphonates for five or more years (and still taking or have since stopped) will be compared with individuals recently starting bisphosphonate treatment and individuals without osteoporosis and not taking bisphosphonates but similar in age. Another cohort of patients who have sustained atypical femur fractures will also be recruited.

Design:

This study will be look at the frequency of subtrochanteric beaking and cortical thickening between three groups of people: long-term users, short-term users, and non-users. Thorough medication usage history, physical examination of the hip and radiographs (x-rays) will be taken three times over the course of three years, and a one time bone density scan will be performed upon enrolling. We will also perform genetic testing for hypophosphatasia in long term asymptomatic users and patients who have sustained the atypical femur fracture.

Outcome measures:

We will be looking for the presence of these "beaks" and measuring the thickness of the hip bone at a certain spot. We are interested in seeing if there is a difference between our three groups of people at first and also if these two features change over three years. We will also monitor for thigh pain, a feature of impending fracture, and if any fractures are found on x-rays. We will compare the prevalence of hypophosphatasia mutations in asymptomatic bisphosphonate users and subjects who have sustained the atypical femur fracture.

ELIGIBILITY:
* INCLUSION CRITERIA - LONGITUDINAL STUDY GROUP:
* For the respective groups, individuals need to be either:

  1. Diagnosis of Osteoporosis or Osteopenia AND have received bisphosphonate therapy for at least 5 years
  2. Diagnosis of Osteoporosis or Osteopenia AND have received bisphosphonate therapy for less than 1 year
  3. Diagnosis of Osteoporosis or Osteopenia AND have received bisphosphonate therapy for 1 to 5 years
  4. No Diagnosis of Osteoporosis or Osteopenia AND have never received bisphosphonate therapy
* Inclusion Criteria In Common Will Be:

  1. Age 50 or older
  2. Ambulatory
  3. Living independently

EXCLUSION CRITERIA - LONGITUDINAL STUDY GROUP:

* Exclusion Criteria Will Be:

  1. Inability to provide informed consent
  2. Cognitive Impairment (MCI/dementia)
  3. Current diagnosis of cancer including: breast, prostate, lung, colon, stomach, bladder, uterus, rectum, thyroid, and kidney
  4. Previous bilateral hip fractures
  5. Pregnancy
  6. Small bowel resections
  7. Malabsorption
  8. Paget s Disease of the Bone
  9. Preexisting osteomalacia, active malignancy, prior bone metastasis, osteogenesis imperfecta, fibrous dysplasia, history of kidney failure.

     INCLUSION CRITERIA - GENETICS STUDY GROUP:

     For the respective groups, individuals need to be either:

  <!-- -->

  1. Diagnosis of atypical femur fracture within the past 10 years, regardless of bisphosphonate use.

     OR
  2. Diagnosis of Osteoporosis or Osteopenia AND have received bisphosphonate therapy for at least 5 years without atypical femur fracture.
* Inclusion Criteria In Common Will Be:

  1. Age 45 or older
  2. Ambulatory
  3. Living independently

     EXCLUSION CRITERIA - GENETICS STUDY GROUP:
* Exclusion Criteria will be:

  1. Inability to provide informed consent
  2. Cognitive Impairment (MCI/dementia)
  3. Current diagnosis of cancer including: breast, prostate, lung, colon, stomach, bladder, uterus, rectum, thyroid, and kidney
  4. Pregnancy
  5. Small bowel resections
  6. Malabsorption
  7. Paget s Disease of the Bone

The following information pertains to individuals in the Longitudinal Group.

Individuals who currently have thigh pain will not be excluded from this study. As the goal of this study is to correlate medication usage with a radiographic feature, individuals concurrently with thigh pain will still be considered, but we will take note of the duration of medication usage and the start of thigh pain per participant history. Duration of thigh pain prior to fracture will likewise be considered. If a current fracture is found on radiographs or suspicion is high for a fracture, selected participants will be sent for MRI of bilateral femurs and participant will be referred back to their primary provider for additional evaluation and treatment.

Individuals who have previously had a unilateral hip fracture or arthroplasty will also not be excluded. As several previous studies have shown, bilateral fractures are not uncommon. We will continue to monitor the progress on the contralateral hip. We will query for details regarding history of first fracture and medication usage. These participants will be subanalyzed for medication usage and time between fractures. Individuals with bilateral (but not unilateral) fractures and bilateral arthroplasty initially will be excluded. However, individuals who are found to have unilateral or bilateral fractures during radiographic studies or undergo unilateral or bilateral arthroplasty during their three years of participation will be allowed to remain in the protocol, and we will assess for change in their anatomy.

Individuals who are being treated with corticosteroids or other types of medications will not be excluded from this study. These variables will be considered confounders and will be analyzed by univariate analysis.

Individuals with anatomical variations such as coxa vara or coxa valga will not be excluded. We will assume that they will be equally distributed into control and treatment groups. These individuals may be at higher risk for atypical fractures, and will be subanalyzed with appropriate femoral-angle matched controls.

Controls that choose to begin bisphosphonate during the study will not be excluded from the study, but will be included in a subanalysis of individuals with less than 3 years of bisphosphonate exposure. Likewise, participants who choose to discontinue bisphosphonate usage will also not be dropped from the study. Analysis will be carried through with groups designated by intent to treat. Users who have taken the drug for 5 years and more who are currently on a drug holiday are eligible (because the drug stays in the bone for so long).

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-05-04; Study Completion 2017-01-11

PRIMARY OUTCOMES:
Difference in prevalence of cortical thickening and beaking between long term users vs. short term or non-users of bisphosphonates.

SECONDARY OUTCOMES:
Difference in rates of cortical thickening over three years between long term users vs. short term or nonusers of bisphosphonates.
Difference in rates of subtrochanteric fractures over three years between long term users vs. short term or nonusers of bisphosphonates.

CONTACTS AND LOCATIONS:
Overall Officials: Michael M Ward, M.D., Principal Investigator — National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS)
Locations (2):
- United States (2):
  - Washington Hospital Center, Washington D.C., District of Columbia
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland

REFERENCES:
- [Background] Shane E, Burr D, Ebeling PR, Abrahamsen B, Adler RA, Brown TD, Cheung AM, Cosman F, Curtis JR, Dell R, Dempster D, Einhorn TA, Genant HK, Geusens P, Klaushofer K, Koval K, Lane JM, McKiernan F, McKinney R, Ng A, Nieves J, O'Keefe R, Papapoulos S, Sen HT, van der Meulen MC, Weinstein RS, Whyte M; American Society for Bone and Mineral Research. Atypical subtrochanteric and diaphyseal femoral fractures: report of a task force of the American Society for Bone and Mineral Research. J Bone Miner Res. 2010 Nov;25(11):2267-94. doi: 10.1002/jbmr.253. PMID 20842676
- [Background] Odvina CV, Zerwekh JE, Rao DS, Maalouf N, Gottschalk FA, Pak CY. Severely suppressed bone turnover: a potential complication of alendronate therapy. J Clin Endocrinol Metab. 2005 Mar;90(3):1294-301. doi: 10.1210/jc.2004-0952. Epub 2004 Dec 14. PMID 15598694
- [Background] Armamento-Villareal R, Napoli N, Panwar V, Novack D. Suppressed bone turnover during alendronate therapy for high-turnover osteoporosis. N Engl J Med. 2006 Nov 9;355(19):2048-50. doi: 10.1056/NEJMc062268. No abstract available. PMID 17093260
- [Derived] Bhattacharyya T, Jha S, Wang H, Kastner DL, Remmers EF. Hypophosphatasia and the risk of atypical femur fractures: a case-control study. BMC Musculoskelet Disord. 2016 Aug 9;17:332. doi: 10.1186/s12891-016-1191-8. PMID 27507156